CLINICAL TRIAL: NCT05364749
Title: Selective Neuroimaging for Head-injured Emergency Patients Who Take Anticoagulant Medication
Brief Title: Selective CT for Anticoagulated Head Injured Patients
Acronym: Can-SCAHn
Status: Recruiting | Type: Observational
Sponsor: Dr. Kerstin de Wit (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Kerstin de Wit, Associate Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: 202104PJ2-461744
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Head Injury; Traumatic Brain Injury; Intracranial Hemorrhage, Traumatic; Blunt Head Injury
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic; Intracranial Hemorrhage, Traumatic; Head Injuries, Closed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal is to derive and a clinical decision rule for safe exclusion of traumatic brain injury without neuroimaging in head-injured ED patients who take anticoagulant medications.

The objectives are to:

1. Derive and externally validate a new highly sensitive and maximally specific clinical decision rule for the exclusion of traumatic brain injury in head-injured ED patients who take anticoagulant medications; and,
2. Estimate the sensitivity and specificity of existing head injury clinical decision rules in head-injured ED patients who take anticoagulant medications.

DETAILED DESCRIPTION:
This is a prospective cohort study enrolling 4000 anticoagulated patients presenting with blunt head trauma to the emergency department. Emergency physicians will record the presence or absence of clinical predictors for traumatic brain injury at the time of assessment. All patients will undergo head CT scanning and are followed for 30 days.

The adjudicated primary outcome is clinically important traumatic brain injury diagnosed at the index ED presentation. The secondary outcome is delayed clinically important traumatic brain injury, diagnosed within 30 days of normal index head CT scan.

The primary analysis will be to derive a novel clinical decision rule which excludes clinically important traumatic brain injury diagnosed at the index ED visit. The secondary analyses will include:

1. The diagnostic accuracy of existing head injury clinical decision rules in diagnosing clinically important traumatic brain injury on index ED visit, in patients who take anticoagulation; and,
2. The sensitivity and specificity of the new and existing rules for the diagnosis of both index and delayed clinically important traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years
* Presents to the emergency department after a head injury
* Patient has a head CT in the emergency department
* Is a current anticoagulant user

Exclusion Criteria:

* Head injury occurred >48 h before patient's arrival to the emergency department
* Penetrating head injury
* Previously enrolled
* Patient resides outside of the hospital's catchment area
* Patient was transferred from another emergency department following neuroimaging
* Patient was not managed by the emergency or trauma physician in the emergency department
* Leaves the emergency department prior to completion of their medical assessment

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolls a anticoagulated emergency department patients presenting within 48 hours of a blunt head injury.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinically important traumatic brain injury | Index emergency department presentation
  Clinically important TBI is defined as the diagnosis of bleeding within the cranial vault, diffuse axonal injury or an isolated skull fracture, which also receives hospital intervention or causes death within 90 days of the traumatic brain injury diagnosis.

SECONDARY OUTCOMES:
Delayed clinically important traumatic brain injury | Diagnosed within 30 days of a negative index head CT scan at the index emergency department presentation
  Clinically important TBI is defined as the diagnosis of bleeding within the cranial vault, diffuse axonal injury or an isolated skull fracture, which also receives hospital intervention or causes death within 90 days of the traumatic brain injury diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin de Wit, MD, Principal Investigator — Queens University
Locations (7):
- Canada (7):
  - University of British Columbia, Vancouver, British Columbia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sinai Health, Toronto, Ontario
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No